CLINICAL TRIAL: NCT01374880
Title: Diagnostic and Prognostic Value of New Biomarkers in Patients With Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); University Paris 7 - Denis Diderot (Other); ThermoFisher Scientific Brahms Biomarkers France (Industry); Hoffmann-La Roche (Industry); Alere San Diego (Industry); Servier (Industry); Helsinki University Central Hospital (Other); University Hospital, Basel, Switzerland (Other); Massachusetts General Hospital (Other); The Cleveland Clinic (Other); Maastricht University Medical Center (Other); Department of Laboratory Medicine, Konventhospital Barmherzige Brueder, Linz, Austria (Unknown); Hospital Universitario Virgen de la Arrixaca (Other); University Hospital Monastir, Tunis (Other); Università degli Studi di Brescia (Other); Intensive and Cardiac Care Unit, Nippon Medical School, Tokyo, Japan (Unknown); Brno University Hospital (Other); University of Cape Town (Other)
Responsible Party: Sponsor
Other Study IDs: CNIL number: 910198; Unité 942 INSERM (Other: CCTIRS number 10.103)
Record Dates: First submitted 2011-04-26; First posted 2011-06-16 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure; Dyspnea; Pulmonary Disease
Keywords: Heart failure; Dyspnea; Heart disease; Pulmonary disease; Natriuretic peptide; Rehabilitation
MeSH Terms: conditions — Heart Failure; Dyspnea; Lung Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers assessment in plasma at different times according to the study cohort.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Dyspnea cohort: Dyspnea cohort
- Stable chronic heart failure: Stable chronic heart failure
- Valvular heart disease: Valvular heart disease
- Ventricular assist device: Ventricular assist device
- Cardiac arrest: Cardiac arrest
- Cardiac rehabilitation: Cardiac rehabilitation

SUMMARY:
The objective of this work is to investigate and then to sequence new biomarkers in the plasma of patients presenting with dyspnea secondary or not to heart failure, and study their diagnostic and prognostic value.

DETAILED DESCRIPTION:
Plasma samples for patients with dyspnea, edema, with or without heart failure; ambulatory or admitted for cardiac decompensation (even with cardiac shock and LVAD) ; or entering a cardiac rehabilitation program, will be prospectively collected.

The objective of this work is to investigate and then to sequence new proteins in the plasma of these patients for diagnostic and prognostic purpose.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with shortness of breath secondary or not to heart failure, even with cardiac shock and LVAD.
* Patients with valvular disease
* chronic stable heart failure.
* post- partum Cardiomyopathy

Exclusion Criteria:

* terminal cancer
* progressive neurological disease
* pregnancy
* opposition of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with dyspnea secondary or not to heart failure. Patients with dyspnea, edema, with heart failure, ambulatory or admitted for cardiac decompensation (even with cardiac shock and LVAD) ; or entering a cardiac rehabilitation program, will be prospectively collected.
  Patients with valvular disease or with chronic heart failure.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-09 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Long term cardiovascular mortality | Prospective at 12 months
  To detect prognostic values of plasma biomarkers, we assess cardiovascular mortality at 3, 6, and 24 months.

SECONDARY OUTCOMES:
Cardiac hospitalization(s) at 3, 6,12 and 24 months | Prospective at 12 months
  We assess cardiac morbidity within 3, 6, and 24 months months after admission
Diagnostic value of new biomarkers. | at day 0
  Assess accuracy of new biomarkers to discriminate heart failure from non-heart failure (negative and positive predictive values)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cohen-Solal, PHD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Lariboisiere hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Badoz M, Arrigo M, Mogenet AC, Sadoune M, Meneveau N, Mebazaa A, Seronde MF. Assessment of successful percutaneous mitral commissurotomy by MRproANP and sCD146. BMC Cardiovasc Disord. 2020 Apr 5;20(1):157. doi: 10.1186/s12872-020-01435-y. PMID 32248819
- [Derived] Van Aelst LNL, Abraham M, Sadoune M, Lefebvre T, Manivet P, Logeart D, Launay JM, Karim Z, Puy H, Cohen-Solal A. Iron status and inflammatory biomarkers in patients with acutely decompensated heart failure: early in-hospital phase and 30-day follow-up. Eur J Heart Fail. 2017 Aug;19(8):1075-1076. doi: 10.1002/ejhf.837. Epub 2017 May 17. No abstract available. PMID 28516737
- [Derived] Vodovar N, Seronde MF, Laribi S, Gayat E, Lassus J, Boukef R, Nouira S, Manivet P, Samuel JL, Logeart D, Ishihara S, Cohen Solal A, Januzzi JL Jr, Richards AM, Launay JM, Mebazaa A; GREAT Network. Post-translational modifications enhance NT-proBNP and BNP production in acute decompensated heart failure. Eur Heart J. 2014 Dec 21;35(48):3434-41. doi: 10.1093/eurheartj/ehu314. Epub 2014 Aug 24. PMID 25157115